CLINICAL TRIAL: NCT04774003
Title: A Placebo-controlled, Participant, Investigator and Sponsor Blinded, Randomized Study to Evaluate the Pharmacokinetics and Pharmacodynamics of Inclisiran Treatment Given as Single Subcutaneous Injection in Chinese Participants With Elevated Low-density Lipoprotein Cholesterol (LDL-C) Despite Treatment With LDL-C Lowering Therapies (ORION-14)
Brief Title: Study of Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Inclisiran in Chinese Participants With Elevated Serum LDL-C
Acronym: ORION-14
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CKJX839A12105
Record Dates: First submitted 2021-02-18; First posted 2021-02-26 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Hyperlipidemia
Keywords: Inclisiran; KJX839; LDL-C; Pharmacokinetics and pharmacodynamics; Chinese participants with elevated serum LDL-C
MeSH Terms: conditions — Hyperlipidemias | interventions — ALN-PCS

STUDY DESIGN:
Intervention Model Description: This is a placebo-controlled study of inclisiran sodium given as a single subcutaneous injection of either 100 mg and 300 mg.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a participant, investigator and sponsor blinded, randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- 300 mg inclisiran sodium (equivalent to 284 mg inclisiran) (Experimental): 300 mg inclisiran sodium (equivalent to 284 mg inclisiran) x 1 dose (n=15) at Day 1
  Interventions: Drug: 300 mg inclisiran sodium (equivalent to 284 mg inclisiran)
- 100 mg inclisiran sodium (equivalent to 94.5 mg inclisiran) (Experimental): 100 mg inclisiran sodium (equivalent to 94.5 mg inclisiran) x 1 dose (n=15) at Day 1
  Interventions: Drug: 100 mg inclisiran sodium (equivalent to 94.5 mg inclisiran)
- Placebo (Placebo Comparator): Placebo x 1 dose (n=10) at Day 1
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 100 mg inclisiran sodium (equivalent to 94.5 mg inclisiran) — 100 mg inclisiran sodium (equivalent to 94.5 mg inclisiran) in 0.5 mL solution. Subcutaneous administration at Day 1
  Other Names: KJX839
  Arms: 100 mg inclisiran sodium (equivalent to 94.5 mg inclisiran)
Drug: Placebo — Inclisiran sodium 0mg (equivalent to inclisiran 0 mg) in 1.5 mL solution. Subcutaneous administration at Day 1
  Arms: Placebo
Drug: 300 mg inclisiran sodium (equivalent to 284 mg inclisiran) — 300 mg inclisiran sodium (equivalent to 284 mg inclisiran) in 1.5 mL solution. Subcutaneous administration at Day 1
  Other Names: KJX839
  Arms: 300 mg inclisiran sodium (equivalent to 284 mg inclisiran)

SUMMARY:
Study to evaluate the pharmacokinetics and pharmacodynamics of inclisiran treatment given as single subcutaneous injection in Chinese participants with elevated low-density lipoprotein cholesterol (LDL-C) despite treatment with LDL-C lowering therapies

DETAILED DESCRIPTION:
The purpose of the study is to characterize pharmacokinetics, pharmacodynamics, safety and tolerability of inclisiran in Chinese participants with elevated serum LDL-C to support inclisiran registration in China.Inclisiran is a long acting RNA therapeutic agent that inhibits the synthesis of PCSK9, leading to reduced circulating LDL-C levels. Three pivotal Phase III studies have been conducted primarily in non-Asian participants to support New Drug Application/Marketing Authorization Application approval of inclisiran globally. This study design is based on the hypothesis that the global inclisiran clinical data primarily obtained in Caucasian participants could be appropriately extrapolated to Chinese participants.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. Male or female participants ≥ 18 years of age at screening
3. Participants should meet fasting serum LDL-C ≥ 100 mg/dL (≥ 2.6 mmol/L) at screening
4. Participants should meet fasting triglyceride < 400 mg/dL (< 4.52 mmol/L) at screening
5. Participants should be receiving a maximally tolerated dose of statin#.
6. For all participants, all the lipid-lowering therapy/ies (such as but not limited to statins and/or ezetimibe) should have remained stable (stable dose and no medication change) for ≥ 30 days before screening with no planned medication or dose change during study participation. #Maximum tolerated dose was defined as the maximum dose of statin that could be taken on a regular basis without intolerable AEs.
7. Participants not receiving statin must have a documented evidence of intolerance to all doses of at least 2 different statins (or the corresponding local definition of complete intolerance to statins)

Exclusion Criteria:

1. Participants diagnosed with any of following: homozygous familial hypercholesterolemia, New York Heart Association class III & IV heart failure, Type 2 diabetes, severe hypertension, active liver disease, HIV infection or any uncontrolled or serious disease;
2. History of drug abuse or unhealthy alcohol use, malignancy of any organ system, or or allergy to the investigational compound/compound class;
3. Major adverse cardiovascular event within 3 months prior to randomization;
4. Calculated glomerular filtration rate ≤30 mL/min by estimated glomerular filtration rate (eGFR) using standardized clinical methodology;
5. Use of other investigational drugs or planned use of other investigational products or devices;
6. Women of child-bearing potential unless they are using basic methods of contraception during dosing of investigational drug (total abstinence, sterilization, barrier methods, hormonal contraception, intrauterine device);
7. Treatment with monoclonal antibodies inhibiting PCSK9 within 90 days prior to screening.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2021-10-18 (Actual); Study Completion 2021-10-18 (Actual)

PRIMARY OUTCOMES:
PK parameters (Cmax) maximum peak observed plasma inclisiran concentration in treated participants | 0-48 hours post-dose
  Pharmacokinetics parameters of inclisiran
PK parameters (Tmax) time to reach maximum peak plasma inclisiran concentration in treated participants | 0-48 hours post-dose
  Pharmacokinetics parameters of inclisiran
PK parameters (T1/2) the elimination half-life associated with the terminal slope of a semi-logarithmic concentration-time curve in inclisiran treated participants | 0-48 hours post-dose
  Pharmacokinetics parameters of inclisiran
PK parameters (AUC) area under the plasma concentration-time curve in inclisiran treated participants | 0-48 hours post-dose
  Pharmacokinetics parameters of inclisiran
Percentage change in Proprotein convertase subtilisin kexin 9 (PCSK9) from baseline overtime | Baseline to Days 5, 8, 15, 30, 60 and 90
  Pharmacodynamics effects of inclisiran
Percentage change in Low density lipoprotein cholesterol (LDL-C) from baseline overtime | Baseline to Days 5, 8, 15, 30, 60 and 90
  Pharmacodynamics effects of inclisiran

SECONDARY OUTCOMES:
Percent change from baseline to Days 30, 60 and 90 in PD parameter Proprotein convertase subtilisin kexin 9 (PCSK9) | Baseline to Days 30, 60 and 90
  Pharmacodynamics differences between inclisiran and placebo
Percent change from baseline to Days 30, 60 and 90 in PD parameter Low density lipoprotein cholesterol (LDL-C) | Baseline to Days 30, 60 and 90
  Pharmacodynamics differences between inclisiran and placebo
Rate of formation of anti-drug antibodies to Inclisiran | Baseline, Days 30 and 90
  Immunogenicity of inclisiran

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- China (3):
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luo Z, Huang Z, Sun F, Guo F, Wang Y, Kao S, Yang G, Huang J, Li J, Zhao S, He Y. The clinical effects of inclisiran, a first-in-class LDL-C lowering siRNA therapy, on the LDL-C levels in Chinese patients with hypercholesterolemia. J Clin Lipidol. 2023 May-Jun;17(3):392-400. doi: 10.1016/j.jacl.2023.04.010. Epub 2023 Apr 29. PMID 37164838
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1308
- See also: Results for CKJX839A12105 from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17979